CLINICAL TRIAL: NCT05784805
Title: Acute Effects of Focused Ultrasound Modulation on EEG Behavior in Status Epilepticus Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Swebilius Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000034504; No NIH funding (Other: 12.06.23)
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Intervention Model Description: Adult patients with ongoing non-convulsive or focal motor SE despite treatment with standard of care antiseizure medications.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with ongoing non-convulsive or focal motor SE (Experimental): Adult patients with ongoing non-convulsive or focal motor SE despite treatment with at least 2 ASMs and who are monitored with surface EEG will be screened and enrolled to receive up to 2 sessions of PLIFU.
  Interventions: Device: PLIFU

INTERVENTIONS:
Device: PLIFU — Participants will be treated with up to 2 sessions of PLIFU (on the same day), while monitored with surface EEG and will be observed for the remainder of the hospital stay as deemed by the primary care team. The system non-invasively delivers ultrasound sonications intracranially that selectively target specific areas of the brain.

SUMMARY:
In this study, the investigators propose Pulsed Low-Intensity Focused Ultrasound (PLIFU) stimulation of brain regions that modulate (thalamus) or generate focal motor seizures (primary motor cortex), with the goal of ameliorating seizure activity in subjects in non-convulsive or focal motor status epilepticus. The course of treatment will consist of an initial 10 minute PLIFU treatment session with an option for a 2nd session if necessary.

The primary objective of this study is to determine whether PLIFU reduces or suppresses epileptic activity in patients with Non-Convulsive Status Epilepticus (NCSE)/Focal Motor Status Epilepticus (FMSE) that have not responded to standard of care.

DETAILED DESCRIPTION:
This study proposes to sonicate epileptic zones or circuits at the bedside with a custom built PLIFU device in two groups of participants experiencing non-convulsive seizures while treated in the Intensive Care Unit (ICU): 1) non-convulsive SE or 2) focal motor Status Epilepticus (SE), targeting the thalami or motor cortical areas responsible for generating ictal activity, respectively.

PLIFU modulation is non-ablative, nonionizing, and noninvasive, while it also preserves the integrity and function of brain tissue. The aim is to quantify ictal and interictal EEG before, during, and after sonication. Experiments will not alter the standard of care and only be implemented after antiseizure medications (ASMs) have been delivered to the patient. PLIFU sonication will be delivered to participants using burst tone and nonthermal parameters for 10 minute exposures.

Hypothesis: PLIFU is a safe and non-invasive treatment that can reduce or suppress epileptic activity.

The pilot data acquired is intended to be used as preliminary data for justifying a larger study.

Recruitment was put on hold from Dec. 2023 to Oct. 2024 due to personnel changes and modifications to study needing approval.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with ongoing NCSE or FMSE despite treatment with at least 2 ASMs
* Provision of signed and dated informed consent form obtained from the next-of-kin/legally authorized representative
* Treated in the ICU while monitored with continuous scalp EEG electrodes

Exclusion Criteria:

* Unable to obtain informed consent
* Presence of an implanted cranial neuromodulation device for treatment of epilepsy
* Pregnancy
* Treatment with another investigational drug or other intervention within 24 hr
* Presence of burr hole(s) or craniotomy
* Subjects with ferromagnetic materials in the head
* Subjects with a TENS unit

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in epileptiform activity | baseline and 10 minutes
  To determine the effect of PLIFU (duration of 10 minutes) on epileptic activity in participants with NCSE/FMSE that have not responded to standard of care using continuous surface EEG. A reduction or suppression of epileptic activity indicates a positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Quraishi, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No